CLINICAL TRIAL: NCT02417480
Title: Differences in Eating Frequency Between Vegan and Omnivorous Diets
Acronym: VeganBytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Clemson University (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Assistant Professor, University of South Carolina
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00043598; 1R21CA187929-01A1 (NIH)
Record Dates: First submitted 2015-04-08; First posted 2015-04-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegan arm (Active Comparator): A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. Researchers will ask participants on a vegan diet to follow their usual diet and exercise habits consistent for the two week study period.
  Interventions: Behavioral: Follow habitual, usual diet
- Omnivorous arm (Experimental): A diet containing all food groups. Researchers will ask participants on an omnivorous diet to follow habitual, usual diet and exercise habits for the first week. During the second week, participants will be asked to switch to a vegan diet for one week and to maintain their usual exercise habits.
  Interventions: Behavioral: Vegan diet; Behavioral: Follow habitual, usual diet

INTERVENTIONS:
Behavioral: Vegan diet — Participants in the omnivorous arm will be asked to follow their normal diet for one week and then follow a vegan diet for one week.
  Arms: Omnivorous arm
Behavioral: Follow habitual, usual diet — Participants will be asked to consume their habitual, usual diet.

SUMMARY:
This study will pilot test the use of two mHealth devices. One is called the Bite Counter and one is called a MisFit. The study will be among a sample of participants (n = 50) to monitor their eating and sleeping habits. The Bite Counter is a wearable watch-like device that detects and records when an individual has taken a bite of food. The benefit of using the Bite Counter is that it places a low-burden on participants to self-monitor their dietary intake. The MisFit is a commercial device that tracks an individual's sleeping and activity.

The purpose of this study is to (1) find out how the Bite Counter calculates daily bites taken on a vegan diet compared to an omnivorous diet, (2) examine differences in sleep and activity between individuals following a vegan diet compared to an omnivorous diet and (3) get feedback from users before the device is tested in larger studies.

DETAILED DESCRIPTION:
In several randomized controlled trials comparing vegan or vegetarian diets to omnivorous dietary approaches, significant weight loss has occurred in the absence of significantly different changes in reported energy intake between groups. This is different than what is seen in studies using traditional weight loss diets (reduced energy omnivorous diets), which demonstrate a greater reduction in energy intake corresponding to greater weight loss. In observational cohort studies, among Adventist Health Study-2 participants following five different diets, BMI was found to be lowest among vegans and highest among omnivores; yet energy intake did not significantly differ among the five groups, averaging 2,000 kcals/day, with the exception of lower energy intake among semi-vegetarians.

This difference in body weight without observed differences in energy intake could possibly be explained by higher levels of physical activity among vegan and vegetarian participants, which have been observed in some of the cohort studies. Physical activity, however, was controlled for in the randomized trials either giving participants identical exercise recommendations, or holding exercise levels constant across experimental groups.

This present study will utilize the Bite Counter to estimate the differences between calories consumed between a vegan diet and an omnivore diet. The significance of using the Bite Counter is that it is a simple way to estimate energy intake. While there are many devices that measure energy expenditure (e.g. various exercise scales and equipment), there are few devices that account for energy intake. Traditional methods of estimating energy intake tend to utilize dietary recalls, but these procedures require much more effort and do not provide real time feedback like the Bite Counter does. Therefore, this study will contribute to current research by capturing data on dietary differences between vegans and omnivores, as well as assessing the usability of this device for dietary self-monitoring. The study will also use an objective physical activity and sleep tracker (the MisFit) to examine differences in exercise and sleeping between omnivorous and vegan participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (18 years and older) that are weight stable individuals (having a BMI between 18.5 - 25
* Participants must have been following their chosen diet for at least the past 6 months
* Participants must be willing to wear a wrist-worn device to track their food intake and physical activity

Exclusion Criteria:

* Participants should have not experienced weight loss or gain ±10 lbs over the past 6 months) and they must not be on a weight loss diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Eating frequency (number of bites taken per day) | 2 weeks
  Number of bites per day will be tracked with a wearable Bite Counter

SECONDARY OUTCOMES:
Energy (kcal) intake | 2 weeks
  Energy intake will be assessed with 24-hour dietary recalls
Physical activity (number of steps/day) | 2 weeks
  Number of steps per day will be assessed with a wrist-worn pedometer (MisFit).
Sleep (number of hours of sleep each night) | 2 weeks
  Number of hours of sleep per night will be assessed with a wrist-word sleep tracking device (MisFit).
Mood (Depression, Anxiety, and Stress Scale (DASS 21) | 2 weeks
  Stress, anxiety, and depression will be assessed with the Depression, Anxiety, and Stress Scale (DASS 21)

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided